CLINICAL TRIAL: NCT06494436
Title: Microvention Aneurysm & Stroke Real-life Data Collection
Acronym: MAESTRO
Status: Recruiting | Type: Observational
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MAESTRO
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Intracranial Aneurysm; Intracranial Aneurysm, Wide Neck Aneurysm, Large Neck Aneurysm Lesion; Aneurysmal Subarachnoid Hemorrhage; Ischemic Stroke; Acute Ischemic Stroke
Keywords: endovascular treatment; stent; flow diverter; hydrocoil; coil; implantable device; FRED; LVIS; WEB; Mechanical Thrombectomy; Aspiration; SOFIA; ERIC; BOBBY
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Cohort 1 will focus on data collection on all Microvention Class III implantable device CE marked used in the treatment of intracranial aneurysms
  Interventions: Device: All Microvention Class III implantable device CE marked
- 2: Cohort 2 will focus on data collection on all Microvention Class III device CE marked used in the treatment of Acute Ischemic Stroke
  Interventions: Device: All Microvention Mechanical Thrombectomy Class III device CE marked

INTERVENTIONS:
Device: All Microvention Class III implantable device CE marked — Endovascular treatment of ruptured or unruptured intracranial aneurysms with commercially available MicroVention implant devices.
  Groups: 1
Device: All Microvention Mechanical Thrombectomy Class III device CE marked — Endovascular treatment of acute ischemic stroke with commercially available MicroVention devices.
  Groups: 2

SUMMARY:
The MAESTRO registry is a post-market, single-arm, non-interventional, multicenter registry

DETAILED DESCRIPTION:
Electronic platform to collect real-world clinical data, evaluate and periodically report safety and effectiveness of CE approved and commercially available Microvention devices used for the endovascular treatment of Intracranial aneurysms and acute ischemic stroke.

ELIGIBILITY:
Inclusion criteria:

* Patient, or another authorized person as per country-specific regulations, is informed of the data collection and gives non-opposition or consent prior to the data collection in accordance with institutional and geographic requirements.
* For Cohort 1, patient is treated for a ruptured or unruptured intracranial aneurysm using a commercially available MicroVention implant device as the primary treatment device and the decision to use this device has been made by the treating physician outside the context of the MAESTRO study.
* For Cohort 2, patient is treated using a commercially available MicroVention mechanical thrombectomy device as the first-line treatment strategy and the decision to use this device has been made by the treating physician outside the context of the MAESTRO study.

Note: For the purposes of this protocol, ancillary/accessory devices such as balloon catheters, carotid stent for extracranial stenosis and other access devices are not considered primary treatment devices. Further, devices used for rescue following attempt of a different primary treatment device are not considered initial primary treatment devices.

Exclusion Criteria:

* Patient is or is expected to be inaccessible for follow-up.
* Patient is participating or intends to participate in another study that changes the site practice.
* Patient is already participating in the MAESTRO study for the same pathology.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Cohort 1: Patients with ruptured or unruptured intracranial aneurysms who are treated endovascularly with commercially available MicroVention implant devices at the direction of the treating physician
  * Cohort 2: Patients with acute ischemic stroke in the cerebral circulation who are treated with mechanical thrombectomy using selected commercially available Microvention devices, at the direction of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Proportion of aneurysms with complete occlusion | 18 (±6) months
  based on Raymond-Roy occlusion classification (RROC) evaluated by an independent Core laboratory
Cohort 2: Proportion of patients achieving final mTICI ≥ 2b revascularization | Mechanical trombectomy Procedure
  based on independent Corelab assessment

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Tomasello, MD, Study Chair — University Hospital Vall D'Hebron; Franziska Dorn, Prof., Study Chair — Bonn University Hospital; Sarah Power, MD, Study Chair — Beaumont Hospital; Krzysztof Kadziolka, MD, Study Chair — John Paul II Independent Public Specialist Western Hospital; Gaultier Marnat, MD, Study Chair — Hôpital Pellegrin, CHU de Bordeaux
Locations (1):
- Álvaro Cunqueiro Hospital - University Hospital Complex of Vigo, Department of Radiology, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No
Confidential document. Only published data will be available